CLINICAL TRIAL: NCT02526394
Title: A Phase III/IV Randomised Open-label Study and Comparison of the Immunogenicity and Safety of a Single Adolescent Booster Dose of a Meningococcal Group C Conjugate-containing Booster Vaccine (Meningitec™, OR NeisVac-C™ , OR Menitorix™), When Given Concurrently With an Acellular Pertussis-containing Booster Vaccine (Repevax™ or IPV-Boostrix™)
Brief Title: Pertussis and Meningitis C Concomitant Vaccination in Adolescents
Acronym: Mutliboost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Multiboost
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2018-04

CONDITIONS: Pertussis; Meningitis; Preventive Immunization; Meningitis; Immunization
MeSH Terms: conditions — Whooping Cough; Meningitis | interventions — Meningococcal Vaccines; Boostrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 (Active Comparator): Repevax + Meningitec
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine
- 2 (Active Comparator): Repevax + Neis-VacC
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine
- 3 (Active Comparator): Repevax + Menitorix
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine
- 4 (Active Comparator): Boostrix + Meningitec
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine
- 5 (Active Comparator): Boostrix + NeisVacC
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine
- 6 (Active Comparator): Boostrix + Menitorix
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine
- 7 (Active Comparator): Repevax + quadrivalent meningococcal conjugate )Nimenrix / Menveo)
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine
- 8 (Active Comparator): Boostrix + quadrivalent meningococcal conjugate )Nimenrix / Menveo)
  Interventions: Biological: Meningococcal vaccine; Drug: Pertussis containing vaccine

INTERVENTIONS:
Biological: Meningococcal vaccine — Meningococcal vaccination
  Other Names: Meningitec, NeisVacC, Menitorix, Menveo, Nimenrix
Drug: Pertussis containing vaccine — Pertussis containing vaccination
  Other Names: Boostrix, Repevax

SUMMARY:
The trial includes groups receiving various combinations of meningitis C and pertussis containing vaccines, to be administered concomitantly in adolescents due their school leaving booster vaccinations (as per UK routine immunisation schedule at 13-17 years of age). Immunogenicity and reactogenicity will be assessed.

DETAILED DESCRIPTION:
Recent numbers of cases of infection with meningococcal C and pertussis (whooping cough), and the characteristics of the people who are these cases, makes it clear that UK adolescents will require booster doses of vaccination for both in the near future. These are increasingly important priorities for the national immunisation policy advisers to the Department of Health, the Joint Committee on Vaccination and Immunisation (JCVI).

There are good indications that the likely target agegroup for these booster vaccinations will be at 14-17 years. Therefore this study seeks primarily to measure antibody responses to the meningitis C and whooping cough vaccines when given at the same time in this agegroup, and see how well the vaccines are tolerated.

Up to 800 adolescents will be recruited across eight study groups. The eight groups arise as a result of combinations of four meningococcal and two whooping cough vaccines each participant will receive a single dose of each of the two types of vaccine (i.e. two injections). Two blood samples will be collected of 10ml each, one prior to vaccination and the second at 35 weeks later. These samples will allow assessment of how the immune system responds to the vaccinations in terms of the antibodies that are present in the blood.

The study will also be assessing how well the vaccines are tolerated in this age group when given together, as described above. Each participant will therefor be asked to complete a health diary for the week following vaccination. This will record any redness/ swelling/ pain at the injection site as well as any illnesses or visits to a GP or hospital.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give written informed consent for participation. If aged below 16 years, parent/legal guardian gives consent while the participant gives written assent for participation in the study.
* Male or female aged 13 years and 6 months (+0 day) to 17 years (+364 days) on the day of consent.
* Completed childhood meningococcal serogroup C and pertussis vaccination according to the UK (catch-up and/or routine) schedule appropriate for the participant's age

Exclusion Criteria:

-

The participant may not enter the study if ANY of the following apply:

* Any contraindication to vaccination as specified in the "Green Book"- Immunisation against Infectious Disease.
* Significant illness including progressive neurological disease or seizure disorder; confirmed or suspected immunosuppressive or immunodeficient conditions; major congenital defects; or known bleeding diathesis (or any condition that may be associated with a prolonged bleeding time).
* Any other significant condition or circumstance which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* History of invasive meningococcal disease or pertussis.
* Significant contact (household or intimate exposure) to an individual with culture proven Neisseria meningitis disease or pertussis in the previous 60 days.
* Received the routine teenage booster dose of tetanus/diphtheria/polio
* Pregnancy

Temporary Exclusion Criteria

* Fever (sublingual temperature ≥ 38°C)
* Received systemic antibiotic(s) (either oral or parenteral) within the past 7 days. For all visits, if allowed by the study visit window, receipt of systemic antibiotics (either oral or parenteral) will delay venepuncture until at least 7 days after cessation of antibiotics.
* Received any blood or blood products within the past 12 weeks.
* Received another investigational agent within 90 days - or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another investigational trial to the end of this study.
* Possibility of pregnancy

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with serogroup C rabbit serum bactericidal assay (rSBA) titres ≥ 8 and ≥ 128 and rSBA geometric mean titre (GMTs) (and percentage with ≥ 4 fold rise compared to baseline). | Day 28 following vaccination
  response to meningococcal vaccination
Pertussis antigen-specific antibody geometric mean concentration (GMCs) in IU/mL for pertussis toxin (PT), Pertactin, and filamentous haemaglutinnin (FHA) and in U/ml for fimbreal antigens (Fims) 2 and 3 | Day 28 following vaccination
  response to pertussis vaccination

SECONDARY OUTCOMES:
Tetanus -specific IgG GMCs in IU/mL and percentages above 0.1 IU/mL | Day 28 following vaccination
  response to tetanus vaccination
Heamophilus type b (Hib)-polyribosylribitol phosphate(PRP)-specific IgG GMCs and proportions achieving IgG concentrations of ≥0.15 or ≥1.00 μg/ml | Day 28 following vaccination
  response to Hib vaccination
Diphtheria-specific IgG GMCs in IU/mL and percentages above 0.1 IU/mL | Day 28 following vaccination
  response to diphtheria vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Gloucestershire primary care, Gloucestershire, Gloucestershire
  - Hertfordshire primary care, Hertfordshire, Hertfordshire